CLINICAL TRIAL: NCT05311020
Title: Efficacy Evaluation of Pitaya Ovule Extract on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH111-REC3-028-2
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-09

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Pitaya Ovule Extract Drink (Experimental)
  Interventions: Dietary Supplement: Pitaya Ovule Extract Drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle per day
  Arms: Placebo drink
Dietary Supplement: Pitaya Ovule Extract Drink — consume 1 bottle per day
  Arms: Pitaya Ovule Extract Drink

SUMMARY:
To assess the efficacy of Pitaya Ovule Extract on skin

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65-year-old males or females

Exclusion Criteria:

* Received medical cosmetic treatment (including cosmetic skin care, laser, fruit acid peeling, injection or plastic surgery, etc.) currently or within one month before the trial
* Outdoor workers (exposed to the sun more than 5 hours a day)
* People who are breastfeeding, pregnant or planning to become pregnant during the test (self-report)
* People with heart, liver, kidney, endocrine and other major organic diseases (self-reported)
* People who have undergone major surgery (according to medical history)
* People who take drugs for a long time
* People with mental illness
* Students who are currently taking courses taught by the principal investigator of this trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
The change of L* (lightness) values | Change from Baseline L* value at 8 weeks
  Spectrophotometer SCM-108 was utilized to measure skin L* value. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® Dual MPA580 was utilized to measure skin elasticity. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Combo Ultrasound module was utilized to measure skin collagen density. Units: arbitrary units
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  IRV skin analyzer was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  IRV skin analyzer was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 8 weeks
  IRV skin analyzer was utilized to measure skin pores. Units: arbitrary units
The change of skin tone | Change from Baseline skin tone at 8 weeks
  IRV skin analyzer was utilized to measure skin tone. Units: arbitrary units
The change of Advanced glycation end products of blood | Change from Baseline AGEs at 8 weeks
  Venous blood was sampled to measure AGEs
The change of RAGE (receptor for advanced glycation end products) of blood | Change from Baseline RAGE at 8 weeks
  Venous blood was sampled to measure RAGE
The change of Matrix metalloproteinases (MMP-2, MMP-9) of blood | Change from Baseline MMPs at 8 weeks
  Venous blood was sampled to measure MMPs

SECONDARY OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Venous blood was sampled to measure renal function biomarkers
The change of fasting blood glucose level | Change from Baseline fasting blood glucose level at 8 weeks
  Venous blood was sampled to measure fasting blood glucose level
Change from Baseline insulin level at 8 weeks | Change from Baseline insulin level at 8 weeks
  Venous blood was sampled to measure insulin level
The change of blood lipid profile | Change from Baseline blood lipid profile at 8 weeks
  Venous blood was sampled to measure blood lipid profile (total cholesterol, HDL-C, LDL-C, triglyceride)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Prof., Principal Investigator — China Medical University, China; Po-Yuan Wu, Dr., Study Director — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taiwan